CLINICAL TRIAL: NCT01295138
Title: Pilot Study of the Effect of Lactulose on Post Caesarean Section Constipation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Fife (Other Government)
Responsible Party: Dr Anthony Davis Consultant Anaesthetist, NHS Fife
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIFEANAES1
Record Dates: First submitted 2010-12-30; First posted 2011-02-14 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2010-12

CONDITIONS: Constipation; Abdominal Pain; Nausea; Vomiting
Keywords: Constipation; Caesarean section; Abdominal Pain; Nausea; Vomiting
MeSH Terms: conditions — Constipation; Abdominal Pain; Nausea; Vomiting | interventions — Lactulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactulose group (Experimental): Group receives 48 hours of lactulose post Caesarean section.
  Interventions: Drug: Lactulose
- Non-lactulose group (No Intervention): Group receives no lactulose post Caesarean section.

INTERVENTIONS:
Drug: Lactulose — Lactulose liquid. 15mls twice daily
  Other Names: Lactugal, Rectulose, Lactulose (non proprietry)
  Arms: Lactulose group

SUMMARY:
Constipation following elective Caesarean sections (CS) is a common problem experienced by up to 50% of patients (1). The causes for this are multifactorial and include manipulation of the bowel during surgery, immobilisation and opiate based anaesthetic and analgesic techniques. To try to alleviate the problem of postoperative constipation, some anaesthetists prescribe postoperative lactulose in addition to postoperative analgesia, although no data exists that shows whether this has any beneficial effect on postoperative constipation.

1. Short term morbidity associated with Caesarean delivery. Hillan EM. Birth. 19 (4): 190-4).

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 16 years or older able to give informed consent undergoing their first or second elective CS

Exclusion Criteria:

* Unable to give informed consent
* A basic level of literacy sufficient to complete postoperative form.
* History of constipation
* Regular opiate use
* Previous bowel surgery or bowel adhesions
* Lactose intolerant
* Diabetic
* Any patient unable to have spinal Anaesthesia
* Allergies/intolerant to bupivacaine, diamorphine, diclofenac, cocodamol, lactulose
* Patients receiving injury to bowel intraoperatively
* Patients receiving additional opiates perioperatively

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-02 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Time in hours to passage of first stool post Caesarean Section. | First 5 days post Caesarean section.
  Time (hours) to first bowel motion post elective LSCS betwwen Lactulose and non-Lactulose groups.

SECONDARY OUTCOMES:
Frequency of abdominal pain between lactulose and non-lactulose groups. | First 5 days post Caesarean section.
  Frequency of abdominal pain between lactulose and non-lactulose groups post Caesarean Section.
Frequency of nausea and vomiting between lactulose and non-lactulose groups | First 5 days post-Caesarean
  Frequency of nausea and vomiting between lactulose and non-lactulose groups post Caesarean Section.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Davis, MBCHB, Principal Investigator — NHS Fife
Locations (1):
- Forth Park Hospital, Kirkcaldy, Fife, United Kingdom